CLINICAL TRIAL: NCT00241150
Title: A Multicenter, Double Blind, Randomized Study With Two Parallel Groups Comparing The Effects Of 12 Weeks Of Treatment With High Dose Valsartan (320 Mg) To Amlodipine On Endothelial Function In Hypertensive Subjects With The Metabolic Syndrome
Brief Title: Diva - The Effects Of 12 Weeks Of Treatment With High Dose Valsartan (320 Mg) To Amlodipine On Endothelial Function In Hypertensive Subjects With The Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A2416
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension; Metabolic Syndrome
Keywords: valsartan; hypertension; metabolic syndrome; endothelial function
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Valsartan

INTERVENTIONS:
Drug: VALSARTAN

SUMMARY:
A STUDY ON WHETHER AN ANTIHYPERTENSIVE MEDICATION PREVENTS DAMAGE TO WALLS OF VEINS IN FEMALE PATIENTS WITH THE METABOLIC SYNDROME (OVERWEIGHT AND OTHER DISORDERS).

ELIGIBILITY:
Inclusion criteria:

Subjects must meet the following inclusion criteria at Visit 1, Visit 2 and Visit 3.

Inclusion criteria for Group A (overweight postmenopausal females with high-normal blood pressure/ mild Stage I hypertension)

1. Non-smoking female outpatients diagnosed as postmenopausal based on age (48 - 65 years) and self-reported absence of menstrual periods for at least one year.
2. Mean blood pressure between 130 - 149 mm Hg systolic and/or 85 - 94 mm Hg diastolic

   • When systolic blood pressure and diastolic blood pressure fall into different categories (high normal versus mild stage I hypertension), the higher category should be selected to classify or group the subject.
3. Body mass index greater than or equal to 26 but less than or equal to 41 kg/m2
4. Subjects who agree not to alter their diet or exercise routine during the study and comply with study specific restrictions 24 hours prior to the next scheduled study visit
5. Subjects who have read, signed and received a copy of the informed consent form prior to the initiation of any study procedures and who agree to participate in all aspects of the study

Exclusion Criteria:

* 1. Non-smoking female outpatients diagnosed as postmenopausal based on age (48 - 65 years) and self-reported absence of menstrual periods for at least one year.

  2. Mean blood pressure between 90 - 129 mm Hg systolic and/or 50 - 84 mm Hg diastolic.

  3. Body mass index greater than or equal to 26 but less than or equal to 41 kg/m2

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline flow-mediated vasodilatation after 12 weeks

SECONDARY OUTCOMES:
Change in baseline brachial artery flow after 12 weeks
Circulating markers of oxidation, inflammation, and fibrinolysis at baseline, 12 weeks
Adverse events and serious adverse events at each study visit for up to 12 weeks
Hematology, blood chemistries, and urine for up to 12 weeks
Vital signs, physical condition, and body weight for up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals